CLINICAL TRIAL: NCT04847518
Title: Effect of Kan-Jang® Supplementation in Patients Diagnosed With COVID-19: A Randomized, Quadruple-blind, Placebo-controlled Trial
Brief Title: Assessment of Efficacy of KAN-JANG® in Mild COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Herbal Institute AB (Industry)
Collaborators: Tbilisi State Medical University (Other); Phytomed AB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHIRD-2021-02; Nr3-2021/87 (Registry Identifier: Registry Identifier: Biomedical Research Ethics Committee)
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a manner of 1:1 for study drug Kan Jang and Standard of Care to Placebo and Standard of Care (Paracetamol)
  The patient study period will last three weeks: active treatment for two weeks and a follow-up period for one week until Hospital discharge to check the side effects and study drug efficacy. During that time, patients will be monitored for adverse events.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomization Sequence of A and B from 1 to 140 will be generated by a qualified pharmacist (QP) at the manufacturing site before the study using a Random number generator. Treatment Randomization Sequence contains information about the distribution of unique random numbers between groups A and B. The QP will keep in secrecy for the clinic, and the investigators the Randomization Sequence and treatment code at the manufacturing site until the study is finalized. Study medications (boxes of placebo and Kan Jang capsules with identical appearance) will be labeled per Treatment Randomization Sequence. It will be provided to an independent statistician for statistical analysis of datasets when all patients complete the treatment. QP will disclose the treatment code providing the information about the actual assignment of treatments A and B to Kan Jang and placebo after statistical analysis of the results of a study where the data obtained from groups A and B will be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kan Jang (Experimental): 70 patients take Kan Jang, two capsules three times a day for the two weeks in the treatment period. Daily dose - 90-120 mg of andrographolides.
  Interventions: Drug: Kan Jang capsules
- Placebo (Placebo Comparator): 70 patients take Placebo, two capsules three times a day for the two weeks in the treatment period
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Drug: Kan Jang capsules — One capsule contains a fixed combination of proprietary
  * Andrographis paniculata Nees. herb, native extract, DER native 4,5-8,0 :1 260 mg (Diterpene lactones andrographolide and 14-deoxy, 11,12- didehydroadnrograholide) 15-20 mg
  * Eleutherococcus senticosus (Rupr. et Maxim) Harms, root, native extract DER native 17-30:1 : 11.4 mg and other inactive excipients (Polycristalline cellulose, Magnesium stearate).
  Other Names: Kan Jang fixed combination
  Arms: Kan Jang
Other: Placebo capsules — Inactive excipients
  Arms: Placebo

SUMMARY:
The complexity of COVID-19 suggests a potential need for a range of therapies, including antiviral agents, immunostimulants, immunosuppressants, adaptogens, and anticoagulants. In this context, implementation of polyvalency drugs, which exhibit a wide range of biological activities and multitarget effects that is common for herbal medicines and specifically for Kan Jang, the fixed combination of Andrographis paniculata (Burm. F.) Wall. ex. Nees and Eleutherococcus senticosus (Rupr. & Maxim.) Maxim which are known to exhibit antiviral, immunomodulatory, and anti-inflammatory effects and clinical efficacy in the respiratory tract of patients with infectious diseases. The purpose of this study is to provide scientific evidence on the effectiveness of Kan Jang for the treatment of mild COVID-19. We hypothesize that Kan Jang will have superior efficacy in amelioration COVID symptoms compared to placebo with a comparable safety profile to placebo. We hypothesize that Kan Jang will increase patients' recovery rate and decrease the duration of illness.

The objective of the study is to assess the efficacy and tolerability of adjuvant treatment with Kan Jang for alleviating the severity of inflammatory symptoms (headache, loss of smell, gustatory dysfunction, rhinorrhea, nasal congestions, cough, sore throat, asthenia, myalgia, and fever) and shortening of their duration in mild COVID-19 patients.

DETAILED DESCRIPTION:
Rationale. Pathogenesis and progression of COVID-19 is a multistep process, which requires correct therapeutic strategy on various steps of initiation of overall defense response to pathogen and its resolution. Consequently, effective treatment of COVID-19 requires pharmaceutical corrections of many components innate, adaptive immune system, phases I-III metabolizing enzymes of detoxifying and repairing systems, and the SARS-Cov-2 virus' life cycle and proliferation.

It can be achieved by multitarget pharmaceutical intervention of herbal preparations with polyvalent and pleiotropic actions on host defense systems, e.g., adaptogens Andrographis paniculata L. (Burm. F.) Wall. ex. Nees and Eleutherococcus senticosus (Rupr. & Maxim.) Maxim, known as natural stress-protective plant extracts that increase adaptability, resilience, and survival of organisms.

A growing body of evidence suggests that extracts of Andrographis paniculata L. (SHA-10) and Eleutherococcus senticosus (SHE-3) are effective and well-tolerated medications for preventing and treating acute viral respiratory infections. WHO recognizes the use of Andrographis paniculata in the symptomatic treatment of upper respiratory infections, bronchitis, and pharyngotonsillitis. Recently, Thailand's health ministry approved using an Herba Andrographidis extract to treat the early stages of Covid-19 as a pilot program amid a flareup in the coronavirus outbreak in Thailand.

The fixed combination of these plants' extracts, the herbal medicinal product Kan Jang®, has been used in Scandinavia for treating symptoms of viral respiratory diseases, such as common colds and influenza, for >30 years. The clinical evidence accumulated indicates that Kan Jang has strong and, in many cases, significant effects on various common cold symptoms. In general, significant improvements were observed in nasal symptoms (e.g., secretion (g/day) frequency, and congestion, throat symptoms (soreness), respiratory problems (incl. cough, frequency of cough), headache, general malaise, fatigue, earache, sleep disturbance, and the objective parameter body temperature and decreased overall total symptoms scores in 5 days of treatment. Furthermore, Kan Jang® sped up patients' recovery and reduced post-influenza complications during the influenza viruses A1 and A3 periods in 1999 and 2000.

Both A. paniculata and E. senticosus and their fixed combination, Kan Jang®, exhibit antiviral, immunomodulatory, and anti-inflammatory effects. Kan Jang® is significantly more effective than the two active ingredients A. paniculata, and E. senticosus extracts alone, presumably due to synergistic interactions in molecular networks deregulated by Kan Jang. A recent study direct antiviral activity of Andrographis, Eleutherococcus, and their combination Kan Jang®, against coronavirus, has been demonstrated: Kan Jang significantly inhibits coronavirus growth in isolated human cells. The antiviral activity of the combinations of Andrographis and Eleutherococcus is more significant than expected. Further studies in COVID-19 patients are warranted to verify whether this observation of the direct antiviral activity of Kan Jang® has clinical significance.

Assessment of primary and secondary endpoints

Treatment benefits will be evaluated by assessment of clinical outcomes, including clinician-reported outcome; observer-reported outcome; performance patient-reported outcomes and biomarkers

Treatment benefits will be evaluated by assessing clinician-, observer- and patient-reported outcomes, including performance outcomes and biomarkers.

Efficacy primary and secondary endpoints will be obtained by intergroup comparison of clinical outcomes changes from baseline during the treatment and follow-up (from Day 1 to Day 14 and day 21 after randomization) in Kan Jang control groups.

A description of the statistical methods to be employed, including the timing of any planned interim analysis (es).

Clinical data at each visit will be recorded using a standardized clinician assessment form and a set of patient rating scales. The data will be entered into an Excel database used as input to statistical software GraphPad (San Diego, CA, USA) Prism software (version 6.03 for Windows), which will be the primary software used for data development and analysis.

Statistical analysis will involve evaluating the patient's change in scores on the test scale from the initial visit (baseline) to intermediate and the final visit and at each scheduled visit of the study. Analysis of changes within treatment groups during the study (Visits 1,2,3 and 4) will be performed by:

* One-way, repeated measures ANOVA (variables with normal distribution),
* Friedman test for repeated several measures (nonparametric data), Results will be calculated using parametric or non-parametric statistical methods depending on the nature of data and applied on intention to treat and per-protocol study groups.

We will evaluate two main questions.

Question 1: was randomization successful, and are groups equal at the beginning of the study?

To assess whether the treatment groups are similar at baseline, we will compare the mean values at baseline for subjects who receive Kan Jang vs. placebo by the Student's parametric independent-measures t-test (variables with normal distribution) or Mann-Whitney non-parametric test, depending on results of normality test.

Question 2: is the effect of Kan Jang treatment superior to the Placebo effect?

Assessment of the efficacy of study medications will be achieved by comparison of mean changes from the baseline (differences before and after treatment of every single patient) between groups using two-way between-within ANOVA in which an interaction effect indicates a different response over time between the two groups and would therefore signal a treatment effect, as well as by multiple comparison t-test (one unpaired test per row),

The primary endpoint is defined as the Duration of the Symptoms. Kaplan-Meier curves will be generated for all endpoints, and medians will be calculated from those curves. The treatment arms will be compared by Mantel-Cox log-rank and Gehan-Breslow-Wilcoxon tests. we will calculate the estimates of treatment hazard ratios based on log-rank tests and 95% CIs.

Intergroup comparison of the number of patients with particular symptoms will be assessed using the odds ratio (OR) statistics of endpoints according to Altman; A/B test of significance of differences of endpoints at 95% confidence, and z-statistic at 95% confidence of statistical significance (Figure 3 b and Supplement 2) (https://www.medcalc.org/calc/odds_ratio.php)

The effect size of the individual and overall symptoms will be calculated as the difference between the effects of Kan Jang and placebo. We will evaluate an overall relative estimate of overall effect size (%) between two treatment groups as.

Effect size (%) = KJ™ - Placebo / KJ™ X 100

We will use a statistical significance level of 5% in the Protocol approved by the health authorities.

We will perform statistical analysis on an intent-to-treat basis.

Safety Analyses

Descriptive statistics (mean, median, standard deviation, minimum, and maximum for continuous variables, and frequencies and percent for categorical variables) will be used to summarize safety measures, which include adverse experiences, physical examination, vital signs, and clinical laboratory tests, etc.

The incidence of adverse events will be compared across treatment groups for descriptive purposes and to identify possible differences in the safety profiles using the odds ratio (OR) statistics of endpoints according to Altman; A/B test of significance of differences of endpoints at 95% confidence; and z-statistic methods for categorical data https://www.medcalc.org/calc/odds_ratio.php.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed (SARS-Cov-2 PCR-positive test) mild COVID-19 infection (in the last three days),
* COVID-19 patient in stable, moderate condition (i.e., not requiring Intensive Care Unit (ICU) admission).
* Subjects must be under observation or admitted to a controlled facility or hospital (home quarantine is not sufficient).
* Able to take medication alone
* Able to give informed consent.

Exclusion Criteria:

* Pulmonary diseases
* Chronic pulmonary diseases
* Chronic rhinosinusitis
* Patient admitted already under invasive mechanical ventilation;
* The patient admitted with the severe acute respiratory syndrome and diagnosed with an etiologic agent other than Covid 19;
* Renal failure requiring dialysis or creatinine ≥ 2.0mg/dl;
* Tube feeding or parenteral nutrition.
* Respiratory decompensation requiring mechanical ventilation.
* Uncontrolled diabetes type 2.
* Hypertension stage 3,
* Autoimmune disease.
* Pregnant or lactating women.
* Patients are taking antibiotics for a reason other than COVID-19 at enrollment.
* Has a chronically weakened immune system (AIDS, lymphoma, chemo-radio- corticosteroid therapy, immunosuppressive pathology);
* Patients treated with chemo-radio-corticosteroid therapy in the last six months.
* Patients with active cancer.
* Taking immunosuppressive drugs (e.g., anti-rejection treatment after organ transplant);
* Already participating in another clinical trial;
* Has any other condition that would prevent safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Duration of symptoms of mild COVID-19: number of days before symptoms disappear | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Time (days) from randomization to symptoms disappear
The severity of the COVID-19 total and individual symptoms: headache, loss of smell, gustatory dysfunction, rhinorrhoea, nasal congestions, cough, sore throat, asthenia, myalgia, and fever | Change from baseline during the period of the treatment and follow up (trough 21 days after randomization)
  Time (days) from randomization to the relief of total and individual mild COVID symptoms scores.
Duration of infection | from Day 1 to Day 14 after randomisation
  Time (days) from randomization to negative SARS-Cov-2 PCR test
Number of participants clinically recovered | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Number of participants (n) without symptoms of mild COVID

SECONDARY OUTCOMES:
Severity of Respiratory symptoms and quality of life scores | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Wisconsin Upper Respiratory Symptom Survey Questionary Score
Cognitive performance test | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  d2-test of attention score
Immune response marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  IL-6 concentration in the serum, pg/ml.
Hypercoagulation marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization
  Dimer-D, ng/ml
Inflammatory marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  C-reactive protein, mg/L
Physical activity | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Assessed by Habitual Physical Activity Questionnaire Score

OTHER OUTCOMES:
Paracetamol intake | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  The number (n) of daily doses (4g) of paracetamol consumed during 14 days from randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Levan Ratiani, PhD, MD, Principal Investigator — The First University Clinic of Tbilisi State Medical University
Locations (1):
- The First University Clinic of Tbilisi State Medical University, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panossian A, Brendler T. The Role of Adaptogens in Prophylaxis and Treatment of Viral Respiratory Infections. Pharmaceuticals (Basel). 2020 Sep 8;13(9):236. doi: 10.3390/ph13090236. PMID 32911682
- [Background] Brendler T, Al-Harrasi A, Bauer R, Gafner S, Hardy ML, Heinrich M, Hosseinzadeh H, Izzo AA, Michaelis M, Nassiri-Asl M, Panossian A, Wasser SP, Williamson EM. Botanical drugs and supplements affecting the immune response in the time of COVID-19: Implications for research and clinical practice. Phytother Res. 2021 Jun;35(6):3013-3031. doi: 10.1002/ptr.7008. Epub 2020 Dec 29. PMID 33373071
- [Background] Panossian A, Seo EJ, Wikman G, Efferth T. Synergy assessment of fixed combinations of Herba Andrographidis and Radix Eleutherococci extracts by transcriptome-wide microarray profiling. Phytomedicine. 2015 Oct 15;22(11):981-92. doi: 10.1016/j.phymed.2015.08.004. Epub 2015 Aug 20. PMID 26407940
- [Background] Panossian A, Seo EJ, Efferth T. Effects of anti-inflammatory and adaptogenic herbal extracts on gene expression of eicosanoids signaling pathways in isolated brain cells. Phytomedicine. 2019 Jul;60:152881. doi: 10.1016/j.phymed.2019.152881. Epub 2019 Mar 10. PMID 30987861
- [Background] Panossian A, Davtyan T, Gukassyan N, Gukasova G, Mamikonyan G, Gabrielian E, Wikman G. Effect of andrographolide and Kan Jang--fixed combination of extract SHA-10 and extract SHE-3--on proliferation of human lymphocytes, production of cytokines and immune activation markers in the whole blood cells culture. Phytomedicine. 2002 Oct;9(7):598-605. doi: 10.1078/094471102321616409. PMID 12487323
- [Background] Panossian A, Wikman G. Efficacy of Andrographis paniculata in upper respiratory tract (URT) infectious diseases and the mechanism of action. In: Evidence and rational based research on Chinese Drugs, Ed. H Wagner and G Ulrich Merzenich (Eds.). Springer Publ. Comp.; 2012. 137-180.